CLINICAL TRIAL: NCT04572516
Title: Topical Application Versus Intra Turbinate Injection of Botulium Toxin Type A In The Treatment of Non Infectious Chronic Rhinosinusitis
Brief Title: Botulium Toxin Type A In Non Infectious Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelalim, MD Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS 3-11-2019
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Chronic rhinosinustitis; Botulium Toxin A
MeSH Terms: conditions — Disease | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical group (Experimental): Topical application in the form of merocel soaked with 20 units of BTX_A (2ml) will be placed at each side of the nasal cavity for 30 minutes.
  Interventions: Drug: BTX A Topical
- Injection group (Experimental): 20 units of BTX_A (2ml) will be injected submucosally in each inferior turbinate using insulin syringe needle after local anesthesia using 10% xylocaine spray .
  Interventions: Drug: BTX A Injection

INTERVENTIONS:
Drug: BTX A Topical — In group A (topical group) ,topical application in the form of merocel soaked with 20 units of BTX_A (2ml) will be placed at each side of the nasal cavity for 30 minutes.
  Other Names: Topical
  Arms: Topical group
Drug: BTX A Injection — In group B (injected group), 20 units of BTX_A(2ml) will be injected submucosally in each inferior turbinate using insulin syringe needle after local anesthesia using 10% xylocaine spray .
  Other Names: Injection
  Arms: Injection group

SUMMARY:
The present work aims to assess the effectiveness and safety of topical application of BTX - A compared with its intra turbinate injection in controlling the symptoms in non infectious chronic rhinosinusitis patients

DETAILED DESCRIPTION:
A prospective comparative study will be carried out on 30 participant of both sex at Otorhinolaryngology Department, Benha University Hospital, it will include patients suffering from non infectious chronic rhinosinustitis symptoms in the form of nasal blockage, rhinorrhea, itching and/or sneezing.

The patients will be divided randomly into two groups:

* Group A (topical group) : 15 patients
* Group B (injected group) : 15 patients

All patients will be subjected to:

1. Full clinical evaluation:

   A) Full history taking B) Clinical examination by
   * anterior rhinoscopy to evaluate the nasal cavity to exclude purulent discharge , nasal polyps or anterior septal deviation.
   * nasal endoscopy to exclude nasal infection signs ,nasal polyps ,the posterior septal deviation or adenoid .

   C) Investigations:CT nose and paranasal sinuses coronal cuts to exclude fungal sinusitis, nasal polyps or other structural abnormalities e.g; posterior septal deviation, conchae bullosa or any other nasal pathology .
2. Intervention :

   * BTX -A available in the Egyptian market in the form of powder vial (Allergan) containing 100 Units, will be dissolved in 10 cc saline to obtain clear colorless solution in which each 1cc contain 10 Units.
   * In group A (topical group) ,topical application in the form of merocel soaked with 20 units of BTX_A (2ml) will be placed at each side of the nasal cavity for 30 minutes.
   * In group B (injected group), 20 units of BTX_A (2ml) will be injected submucosally in each inferior turbinate using insulin syringe needle after local anesthesia using 10% xylocaine spray .
3. Follow Up Follow up visits will be at 1,2,4,6,8 weeks, patients will be assessed and questionnaired about severity of the symptoms and possible adverse effects including epistaxis and nasal dryness .

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent symptoms of chronic non infectious rhinosinusitis not responding to previous lines of treatment including antihistaminics ,nasal decongestant, and or nasal steroid spray will be included in this study.

Exclusion Criteria:

* Patients with major structural deformities(septal deviation , adenoid hypertrophy, nasal valve pathology or nasal polyps).
* Having systemic illness such as DM, HTN, Malignancy or Tuberculosis.
* History of nasal surgery such as turbinate reduction surgery orseptoplasty.
* Acute rhinosinusitis findings; e.g purulent or mucopurulent nasal discharge
* Radiological finding of nasal tumors or fungal sinusitis.
* Any accompanying disease such as glaucoma or prostate hypertrophy or myasthenia that might be aggravated by anticholinergic therapy .
* use of systemic or local corticosteroid less than 1 month prior the study.
* Pregnancy or lactation.
* History of allergy to botox or local anesthetic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
the rhinitis symptom severity | 2 months
  the rhinitis symptom severity questionnaire, this is questionnaire consists of 4 items (nasal obstruction, rhinorrhea , sneezing and or nasal itching) . each symptom given score from 0 to 3 ( 0 = none, 1 = mild, 2 = moderate and 3 = severe)

SECONDARY OUTCOMES:
possible adverse effects | 2 months
  epistaxis and nasal dryness (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman A Abdelalim, MD, Principal Investigator — Benha University; Mohamed A Elsayed, MD, Study Chair — Benha University; Naslshah G Kazeem, MD, Study Chair — Benha University; Aya L Hassan, Resident, Study Chair — Benha University
Locations (1):
- Benha University Hospital, Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang EZ, Tan S, Loh I. Botolinum toxin in rhinitis: Literature review and posterior nasal injection in allergic rhinitis. Laryngoscope. 2017 Nov;127(11):2447-2454. doi: 10.1002/lary.26616. Epub 2017 Jul 6. PMID 28681969
- [Background] Ozcan C, Vayisoglu Y, Dogu O, Gorur K. The effect of intranasal injection of botulinum toxin A on the symptoms of vasomotor rhinitis. Am J Otolaryngol. 2006 Sep-Oct;27(5):314-8. doi: 10.1016/j.amjoto.2006.01.008. PMID 16935174